CLINICAL TRIAL: NCT06041477
Title: A Randomized Controlled Study of the Efficacy of Hepatic Arterial Perfusion Chemotherapy Concurrently Compared to Sequentially Combined With Targeted and Immunotherapy in Potentially Resectable Intermediate and Advanced HCC
Brief Title: Concurrently vs Sequentially Combined HAIC With Targeted and Immunotherapy in Potentially Resectable HCC
Acronym: HAIC
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Collaborators: The First Affiliated Hospital, Guangzhou University of Traditional Chinese Medicine (Other); Affiliated Hospital of Guangdong Medical University (Other); First People's Hospital of Foshan (Other)
Responsible Party: Principal Investigator, Wei Wei, Professor, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SL-B2022-793-01; 2023001 (Other: SUN Yat-sen University)
Record Dates: First submitted 2023-07-23; First posted 2023-09-18 (Actual); Last update posted 2024-08-27 (Actual); Status verified 2024-08

CONDITIONS: Hepatocellular Carcinoma; Chemotherapy Effect; Chemotherapeutic Toxicity
Keywords: Hepatic artery infusion chemotherapy; Tyrosine kinase inhibitors; Immune checkpoint inhibitors; Intermediate and advanced stage hepatocellular carcinoma; combined therapy; conversion resection
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Oxaliplatin; Leucovorin; Fluorouracil

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- concurrent treatment group (Experimental): Participants receive two cycles of HAIC (the drugs are oxaliplatin 135mg/m2 over 3hrs, calcium folinic acid 400mg/m2 or levofolinic acid 200mg/ m2 over 1.5hrs, 5-FU 400mg/m2 over 2hrs, 5-FU 2400mg/m2 over 46hrs,every 4 weeks) in combination with targeted drug (lenvatinib 8mg/day) and immunotherapy (PD-1 antibody, dosage and frequency according to instructions), then evaluate the response of tumor, those who achieve complete response (CR) will receive surgical resection or follow-up, those with partial response (PR) or stable disease (SD) continue two cycles of combined therapy, and those with progress disease (PD) will be withdrawn and receive other treatments. After four cycles of combined therapy, second evaluation of efficacy will be performed, those who achieve CR will receive surgical resection or follow-up observation, and the other patients will be evaluated for the possibility of surgical resection or the subsequent treatment.
  Interventions: Drug: Oxaliplatin,calcium folinic acid, levofolinic acid, 5-FU; Drug: Concurrent Lenvatinib; Drug: Concurrent PD-1 antibody
- sequential treatment group (Active Comparator): Participants receive two cycles of HAIC (drugs of oxaliplatin 135 mg/m2 over 3 hours; calcium folinic acid 400 mg/m2 or levofolinic acid 200 mg/m2 over 1. 5 hours, 5-FU 400 mg/m2 over 2 hours, and 5-FU 2400 mg/m2 over 46 hours,every 4 weeks), then evaluate the response of tumor, and those who achieve complete response (CR ) will receive surgical resection or follow-up, while other patients continue to receive two cycles of combination therapy, i.e. HAIC combined with targeted drug (levatinib 8mg/day) and immunotherapy (PD-1 antibody, dose and frequency according to instructions). After four cycles, a second efficacy assessment will be performed, and patients who achieve CR will undergo surgical resection or follow-up observation, and the other patients will be evaluated for the possibility of surgical resection or the subsequent treatment.
  Interventions: Drug: Oxaliplatin,calcium folinic acid, levofolinic acid, 5-FU; Drug: Sequential Lenvatinib; Drug: Sequential PD-1 antibody

INTERVENTIONS:
Drug: Oxaliplatin,calcium folinic acid, levofolinic acid, 5-FU — Hepatic arterial infusion chemotherapy with (oxaliplatin 135mg/m2 over 3hrs, calcium folinic acid 400mg/m2 or levofolinic acid 200mg/ m2 over 1.5hrs, 5-FU 400mg/m2 over 2hrs, 5-FU 2400mg/m2 over 46hrs,every 4 weeks)
  Other Names: Hepatic arterial infusion chemotherapy (HAIC)
Drug: Concurrent Lenvatinib — Lenvatinib 8mg/day combined with the HAIC from the first cycle
  Other Names: Concurrent targeted therapy
  Arms: concurrent treatment group
Drug: Concurrent PD-1 antibody — PD-1 antibody which is approved by authorities for HCC treatment combined with the HAIC from the first cycle (dosage and frequency according to instructions)
  Other Names: Concurrent immunotherapy
  Arms: concurrent treatment group
Drug: Sequential Lenvatinib — Lenvatinib 8mg/day combined with the HAIC from the third cycle for those patients who do not achieve complete response (CR)
  Other Names: Sequential targeted therapy
  Arms: sequential treatment group
Drug: Sequential PD-1 antibody — PD-1 antibody which is approved by authorities for HCC treatment combined with the HAIC from the third cycle for those patients who do not achieve complete response (CR) (dosage and frequency according to instructions)
  Other Names: Sequential immunotherapy
  Arms: sequential treatment group

SUMMARY:
The goal of this clinical trial is to compare HAIC concurrently with sequentially combined with targeted and immunotherapies in terms of efficacy and safety in patients with potentially resectable intermediate and advanced HCC (CNLC stage IIa~IIIa). The main questions it aims to answer are:

* Does a "strong combination" regimen of three simultaneous treatments (HAIC, targeted agents and immunotherapy) definitely result in a higher surgical conversion rate and better survival benefit?
* Can the combination of targeted and immunotherapies based on patients' response to HAIC therapy avoid over-treatment of some patients without affecting the surgical conversion rate and overall survival? Participants will be randomly assigned to receive either HAIC concurrently or sequentially combined with targeted and immunotherapies.

Researchers will compare concurrent treatment group with sequential treatment group to see if there are different in terms of the conversion resection rate, long-term survival, and safety.

DETAILED DESCRIPTION:
Participants in the concurrent treatment group will receive two cycles of HAIC (the drugs are oxaliplatin 135mg/m2 over 3hrs, calcium folinic acid 400mg/m2 or levofolinic acid 200mg/ m2 over 1.5hrs, 5-FU 400mg/m2 over 2hrs, 5-FU 2400mg/m2 over 46hrs,every 4 weeks) in combination with targeted drug (lenvatinib 8mg/day) and immunotherapy (PD-1 antibody, dosage and frequency according to instructions), then evaluate the response of tumor, those who achieve complete response (CR) will receive surgical resection or follow-up, those with partial response (PR) or stable disease (SD) continue two cycles of combined therapy, and those with progress disease (PD) will be withdrawn and receive other treatments. After four cycles of combined therapy, second evaluation of efficacy will be performed, those who achieve CR will receive surgical resection or follow-up observation, and the other patients will be evaluated for the possibility of surgical resection or the subsequent treatment.

Participants in the sequential treatment group will receive two cycles of HAIC (drugs of oxaliplatin 135 mg/m2 over 3 hours; calcium folinic acid 400 mg/m2 or levofolinic acid 200 mg/m2 over 1. 5 hours, 5-FU 400 mg/m2 over 2 hours, and 5-FU 2400 mg/m2 over 46 hours,every 4 weeks), then evaluate the response of tumor, and those who achieve complete response (CR ) will receive surgical resection or follow-up, while other patients continue to receive two cycles of combination therapy, i.e. HAIC combined with targeted drug (levatinib 8mg/day) and immunotherapy (PD-1 antibody, dose and frequency according to instructions). After four cycles, a second efficacy assessment will be performed, and patients who achieve CR will undergo surgical resection or follow-up observation, and the other patients will be evaluated for the possibility of surgical resection or the subsequent treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 and ≤75 years;
2. ECOG PS score of 0~1;
3. Clinical or pathological diagnosis of hepatocellular carcinoma and meeting the stage IIa-IIIa of CNLC staging according to the relevant definitions in the 2015 edition of the Guidelines for Standardized Pathological Diagnosis of Primary Liver Cancer;
4. Not having received previous treatment against hepatocellular carcinoma;
5. Those who cannot be surgically resected after discussion by the multidisciplinary team of the participating centers , but have a potential chance of resection after conversion therapy, including: multiple tumors located in one lobe of the liver; portal vein cancer thrombus not reaching the main trunk, which can be resected together with the primary focus;
6. Laboratory tests meet the following conditions, or the following conditions can be achieved with short-term treatment:

   Neutrophil count ≥2.0×109/L; Hemoglobin ≥ 100 g/L; Platelet count ≥ 75 × 109/L; Plasma albumin level ≥ 35 g/L; Plasma total bilirubin less than 2 times the upper limit of normal; Plasma alanine aminotransferase (ALT) less than 3 times the upper limit of normal; Plasma aspartate aminotransferase (AST) less than 3 times the upper limit of normal; Plasma creatinine less than 1.5 times the upper limit of normal; Plasma prothrombin time is normal or exceeds the upper limit of normal value by ≤ 4 seconds; Prothrombinogen international normalized ratio (INR) ≤ 2.2;
7. Patients were fully informed about the study and signed an informed consent form.

Exclusion Criteria:

1. Those with severe comorbidity including cardiac, cerebral, pulmonary, renal, and other vital organ function damage, combined with severe infections or other serious concomitant diseases (> grade 2 CTCAE Version 5.0 adverse events), who cannot tolerate the treatment;
2. Those with a history of other malignant tumors;
3. Those with a history of related drug allergy;
4. Those with known hypersensitivity to any component of the targeted and immunologic drugs to be applied;
5. Those with a history of organ transplantation;
6. Those who have received previous treatment targeting hepatocellular carcinoma (including interferon);
7. Those with co-infection with HIV;
8. Those with drugs abuse;
9. Those who have had gastrointestinal bleeding or cardiovascular events within the last 30 days;
10. Pregnant or breastfeeding women, or women of childbearing age who do not wish to use contraception;
11. Persons with concomitant psychiatric disorders that preclude informed consent or affect acceptance of treatment;
12. Other factors that may affect patient enrollment and assessment results.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 540 (Estimated)
Dates: Start 2023-10-31 (Actual); Primary Completion 2027-07 (Estimated); Study Completion 2030-07 (Estimated)

PRIMARY OUTCOMES:
OS | From date of randomization until the date of death from any cause, assessed at least 36 months
  Overall survival of the participants

SECONDARY OUTCOMES:
PFS | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed at least 36 months
  Progression-free survival of the participants
ORR | Assessed at the end of Cycle 2 and Cycle 4 (each cycle is 28 days)
  Objective response rates, which means the proportion of patients with efficacy assessment of complete response and partial response for the size of intrahepatic target lesions according to mRECIST criteria and RECIST v1.1 criteria respectively.
DCR | Assessed at the end of Cycle 2 and Cycle 4 (each cycle is 28 days)
  Disease control rates, which means the proportion of patients with efficacy assessment of complete response, partial response and stable disease for the size of intrahepatic target lesions according to mRECIST criteria and RECIST v1.1 criteria respectively.
CRR | This outcome measure will be assessed at the end of Cycle 4 (each cycle is 28 days)
  Conversion resection rate refer to the proportion of patients in both groups who actually underwent subsequent surgical resection.
Safety profiles of all participants | This outcome measure will be assessed at the end of Cycle 1 to 4(each cycle is 28 days), and every 3 months through study completion, an average of 3 years
  Adverse Events and Severe Adverse Events evaluated based on Common Terminology Criteria for Adverse Events (CTCAE) Version 5.0

CONTACTS AND LOCATIONS:
Overall Officials: Wei Wei, Ph.D, M,D, Principal Investigator — Sun Yat-sen University
Locations (1):
- SUN Yat-sen University Cancer Center, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No
From the perspective of protecting the privacy of participants, there was no participant data (IPD) plan in this study.

REFERENCES:
- [Result] Sung H, Ferlay J, Siegel RL, Laversanne M, Soerjomataram I, Jemal A, Bray F. Global Cancer Statistics 2020: GLOBOCAN Estimates of Incidence and Mortality Worldwide for 36 Cancers in 185 Countries. CA Cancer J Clin. 2021 May;71(3):209-249. doi: 10.3322/caac.21660. Epub 2021 Feb 4. PMID 33538338
- [Result] Park JW, Chen M, Colombo M, Roberts LR, Schwartz M, Chen PJ, Kudo M, Johnson P, Wagner S, Orsini LS, Sherman M. Global patterns of hepatocellular carcinoma management from diagnosis to death: the BRIDGE Study. Liver Int. 2015 Sep;35(9):2155-66. doi: 10.1111/liv.12818. Epub 2015 Mar 25. PMID 25752327
- [Result] Forner A, Reig M, Bruix J. Hepatocellular carcinoma. Lancet. 2018 Mar 31;391(10127):1301-1314. doi: 10.1016/S0140-6736(18)30010-2. Epub 2018 Jan 5. PMID 29307467
- [Result] Schwartz JD, Schwartz M, Mandeli J, Sung M. Neoadjuvant and adjuvant therapy for resectable hepatocellular carcinoma: review of the randomised clinical trials. Lancet Oncol. 2002 Oct;3(10):593-603. doi: 10.1016/s1470-2045(02)00873-2. PMID 12372721
- [Result] Shi HY, Wang SN, Wang SC, Chuang SC, Chen CM, Lee KT. Preoperative transarterial chemoembolization and resection for hepatocellular carcinoma: a nationwide Taiwan database analysis of long-term outcome predictors. J Surg Oncol. 2014 Apr;109(5):487-93. doi: 10.1002/jso.23521. Epub 2013 Nov 30. PMID 24293372
- [Result] He M, Li Q, Zou R, Shen J, Fang W, Tan G, Zhou Y, Wu X, Xu L, Wei W, Le Y, Zhou Z, Zhao M, Guo Y, Guo R, Chen M, Shi M. Sorafenib Plus Hepatic Arterial Infusion of Oxaliplatin, Fluorouracil, and Leucovorin vs Sorafenib Alone for Hepatocellular Carcinoma With Portal Vein Invasion: A Randomized Clinical Trial. JAMA Oncol. 2019 Jul 1;5(7):953-960. doi: 10.1001/jamaoncol.2019.0250. PMID 31070690
- [Result] Lyu N, Kong Y, Mu L, Lin Y, Li J, Liu Y, Zhang Z, Zheng L, Deng H, Li S, Xie Q, Guo R, Shi M, Xu L, Cai X, Wu P, Zhao M. Hepatic arterial infusion of oxaliplatin plus fluorouracil/leucovorin vs. sorafenib for advanced hepatocellular carcinoma. J Hepatol. 2018 Jul;69(1):60-69. doi: 10.1016/j.jhep.2018.02.008. Epub 2018 Feb 20. PMID 29471013
- [Result] He MK, Le Y, Li QJ, Yu ZS, Li SH, Wei W, Guo RP, Shi M. Hepatic artery infusion chemotherapy using mFOLFOX versus transarterial chemoembolization for massive unresectable hepatocellular carcinoma: a prospective non-randomized study. Chin J Cancer. 2017 Oct 23;36(1):83. doi: 10.1186/s40880-017-0251-2. PMID 29061175
- [Result] Li S, Mei J, Wang Q, Guo Z, Lu L, Ling Y, Xu L, Chen M, Zheng L, Lin W, Zou J, Wen Y, Wei W, Guo R. Postoperative Adjuvant Transarterial Infusion Chemotherapy with FOLFOX Could Improve Outcomes of Hepatocellular Carcinoma Patients with Microvascular Invasion: A Preliminary Report of a Phase III, Randomized Controlled Clinical Trial. Ann Surg Oncol. 2020 Dec;27(13):5183-5190. doi: 10.1245/s10434-020-08601-8. Epub 2020 May 16. PMID 32418078
- [Result] Li SH, Mei J, Cheng Y, Li Q, Wang QX, Fang CK, Lei QC, Huang HK, Cao MR, Luo R, Deng JD, Jiang YC, Zhao RC, Lu LH, Zou JW, Deng M, Lin WP, Guan RG, Wen YH, Li JB, Zheng L, Guo ZX, Ling YH, Chen HW, Zhong C, Wei W, Guo RP. Postoperative Adjuvant Hepatic Arterial Infusion Chemotherapy With FOLFOX in Hepatocellular Carcinoma With Microvascular Invasion: A Multicenter, Phase III, Randomized Study. J Clin Oncol. 2023 Apr 1;41(10):1898-1908. doi: 10.1200/JCO.22.01142. Epub 2022 Dec 16. PMID 36525610